CLINICAL TRIAL: NCT02644421
Title: Phase Ib Randomized, Double-Blind, Latin Square Crossover, Clinical Trial to Evaluate the Safety and Analgesic Efficacy of VVZ-149 v. Lidocaine v. Placebo in Lumbar Radiculopathy
Brief Title: Clinical Trial to Evaluate the Safety and Analgesic Efficacy of VVZ-149 in Lumbar Radiculopathy (Sciatica)
Acronym: LMR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Christine N. Sang, MD, MPH, Director, Translational Pain Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-P-002050
Record Dates: First submitted 2015-12-08; First posted 2015-12-31 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Radiculopathy; Sciatica
Keywords: Neuropathic Pain; Sciatica
MeSH Terms: conditions — Radiculopathy; Sciatica; Neuralgia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VVZ-149 (Experimental): The following doses will be administered intravenously:
  * Loading Dose: 1.8 mg/kg VVZ-149 over 0.5 hours
  * Maintenance infusion: 1.3 mg/kg/hr VVZ-149 over 7.5 hours
  Interventions: Drug: VVZ-149
- Lidocaine (Active Comparator): The following doses will be administered intravenously:
  * Lidocaine 4mg/kg LBM over 0.5 hours
  * Normal saline over 7.5 hours
  Interventions: Drug: Lidocaine
- Placebo (Placebo Comparator): Normal saline administered intravenously over 8 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VVZ-149
  Arms: VVZ-149
Drug: Lidocaine
  Arms: Lidocaine
Drug: Placebo
  Arms: Placebo

SUMMARY:
Double-blind, crossover, randomized, 3x3 Latin square, placebo-controlled study of single intravenous dose administration of VVZ-149. To demonstrate assay sensitivity, lidocaine will be administered as a positive control. The study will take place during a single inpatient visit involving three separate treatment periods, each with a washout of (>16-hours. Study drugs (VVZ-149 vs. lidocaine vs. normal saline, NS) will be administered intravenously.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have a history of persistent pain secondary to unilateral monoradiculopathy present for a minimum of 3 months prior to the study, with an average pain intensity score of at least moderate over at least 50% of the day for the 7 days prior to the screening visit and over the 7 days prior to starting study medication.
2. Males or females between 18 and 70 years of age, inclusive. Females who are pregnant or breastfeeding will be excluded from the trial.
3. Subjects must be in generally good health, either using no medication or using a stabilized medication regimen for chronic and well-controlled conditions such as hypertension, allergies, stable endocrinopathies (e.g. hypothyroidism), etc. Subjects with other active diseases will be reviewed on a case-by-case basis by the principal investigator.
4. No concomitant therapy with any medication that is a known significant inhibitor or inducer of CYP450 2D6 and CYP3A4, at the discretion of the PI.
5. Normal or clinically insignificant screening laboratory tests:

   * Serum BUN, creatinine, bicarbonate, calcium, chloride, potassium, sodium, lactate dehydrogenase, inorganic phosphate, total protein, glucose, albumin, and uric acid. WBC, absolute neutrophil count, hemoglobin, hematocrit, and platelets. SGOT (AST), SGPT (ALT), total bilirubin, alkaline phosphatase, TSH/T4, urinalysis, and urine toxicology screen.
   * Electrocardiogram (12-lead). Any significant laboratory abnormalities will be reviewed by the principal investigator prior to inclusion of the subject in the study.
6. Willingness to restrict analgesic therapy during inpatient admission days to the allowed rescue analgesic agent permitted by the study (acetaminophen).
7. Subjects must have normal cognitive function and communicative ability in the English language.
8. Subjects must be able to provide meaningful written informed consent.
9. Subjects must be able to maintain complete required questionnaires, and must be able to fulfill all other conditions of the protocol.

Exclusion Criteria:

1. Female subjects who are pregnant or breastfeeding, or plan to become pregnant while participating in the study.
2. Subjects with a previous history of multiple or severe drug allergies, including lidocaine.
3. Subjects with a history of or current chronic substance abuse, including alcohol.
4. Subjects who have participated in a study of an investigational drug or device within 30 days prior to screening for this study. Subjects must agree not to participate in other investigational drug or device studies during the entire course of this study (beginning with the screening visit).
5. Subjects with the following abnormal clinical evaluations:

   * Impaired renal function defined as BUN > 45 or creatinine >2.0 and/or impaired liver function defined as liver transaminases, alkaline phosphatase, or bilirubin greater than 1.5 x upper limit of normal laboratory values.
   * Prolonged PR (>200 ms) interval on electrocardiogram (12-lead). Subjects presenting with the above laboratory abnormalities may be allowed on a case-by-case basis at the discretion of the principal investigator.
6. Subjects who intend to donate blood or blood products while participating in this study, and for 30 days following completion of the study.
7. Subjects with clinically significant renal, hepatic, or cardiac disease, with seizure disorders, or with a clinical history of life-threatening arrhythmias (i.e. torsades de pointes).
8. Subjects with a severe neuropsychiatric disorder requiring treatment.
9. Subjects with sensitivity to amide-type local anesthetics.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2015-11; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Number of subjects with treatment-related Adverse Events as assessed using an internal, categorical severity/relationship scale | over 8 hour infusion
  The number of subjects who report mild, moderate or severe treatment-emergent adverse events that are deemed by the investigator to be possibly, probably, or definitely related to the study medication

SECONDARY OUTCOMES:
Reduction in Pain Intensity using the 11-pt Likert Pain Intensity Scale | over 8 hour infusion
  Reductions in pain intensity from baseline will be calculated using data obtained over the 8 hour infusion from the 11-pt Likert Pain Intensity Scale

CONTACTS AND LOCATIONS:
Overall Officials: Christine N Sang, MD MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Translational Pain Research, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No